CLINICAL TRIAL: NCT06524310
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Cognitive Functions and Behavior in Individuals With Autism Spectrum Disorder ( ASD)
Brief Title: Effects of rTMS on Cognitive Functions and Behavior in Individuals With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Hayfa Ali Alghabban, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: rTMS_ASD_SA
Record Dates: First submitted 2024-06-30; First posted 2024-07-29 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD, Autism Spectrum Disorder; Repetitive Transcranial Magnetic Stimulation , rTMS; Cognitive function; Social cognition; autistic behaviors; social interaction; sensory problems; excitation to inhibition imbalance; glutamate excitotoxicity
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with a waiting list control design.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the waiting list control design, blinding of participants and their guardians to group allocation was not possible. However, the clinicians performing the outcome assessments were blinded to the participants' group assignments to minimize potential observer bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- active rTMS group (Experimental): Male and female ASD individuals aged between 5 and 11 years old who have been diagnosed with ASD. They should have a confirmed clinical diagnosis according to the DSM-5. This will be verified by a diagnostic report or direct communication with the diagnosing clinician. Also, with normal hearing based on past hearing screens. Exclusion criteria to ensure participant safety for the rTMS intervention and included: (1) a history of seizures or epileptiform activity; (2) the presence of any metallic implants within the cranium; (3) a history of significant head trauma or loss of consciousness; and (4) the presence of implanted electronic medical devices (e.g., pacemakers, cochlear implants). All participants in both study groups did not stop their medical or behavioral therapy for ASD. However, participants will be instructed to have a consistent medication regimen or behavioral treatment for at least one month before enrollment and throughout the trial.
  Interventions: Device: Stimulation with low frequency rTMS at 1 Hz
- wait-list-control group (No Intervention): Male and female ASD individuals aged between 5 and 11 years old who have been diagnosed with ASD. They should have a confirmed clinical diagnosis according to the DSM-5. This will be verified by a diagnostic report or direct communication with the diagnosing clinician. Also, with normal hearing based on past hearing screens. Exclusion criteria to ensure participant safety for the rTMS intervention and included: (1) a history of seizures or epileptiform activity; (2) the presence of any metallic implants within the cranium; (3) a history of significant head trauma or loss of consciousness; and (4) the presence of implanted electronic medical devices (e.g., pacemakers, cochlear implants). All participants in both study groups did not stop their medical or behavioral therapy for ASD. However, participants will be instructed to have a consistent medication regimen or behavioral treatment for at least one month before enrollment and throughout the trial.

INTERVENTIONS:
Device: Stimulation with low frequency rTMS at 1 Hz — Stimulation with low-frequency rTMS at 1 Hz with 90% MT will be applied with a total of 180 pulses each time, which contains 18 trains with ten pulses and an interval of 20 s between any two adjacent trains. The TMS treatment course will be administered twice per week for 9 weeks; the first six treatments will be over the left DLPFC, the second six sessions will be over the right DLPFC, and the remaining six sessions will be placed on the bilateral DLPFC stimulation.
  Other Names: NeuroStar TMS Therapy System (Neuronetics, Inc; Malvern, Pennsylvania). with figure of 8- Coil and a special sensory guard ( SenStarTreatment Link).
  Arms: active rTMS group

SUMMARY:
Autism spectrum disorder (ASD) is a complex neurodevelopmental disorder with core symptoms that include impairments in social communication and restricted and repetitive behaviors, interests, and activities. Social cognition is a broad term used to understand, perceive, and interpret information about others and ourselves in a social context. Impairments in social cognition are often highlighted as a potential mechanism underlying social disability in autism spectrum disorder. Repetitive transcranial magnetic stimulation is a noninvasive technique that modulates brain activity through targeted electromagnetic pulses. It's one of the methods used to deliver electrical stimuli through the scalp in conscious humans. Recently, rTMS has not only been used for the treatment of major depressive disorders, but it has also been advanced as a potential therapeutic technique to treat neurologic disorders such as Parkinson's disease, Huntington's disease, amyotrophic lateral sclerosis, and multiple sclerosis, and many other neuropsychiatric disorders. High-order cognitive functions, such as Executive function (EF) and social cognition, rely on neural network oscillations in the gamma frequency (30-80 Hz) band. It has been proposed that GABA-inhibitory interneurons in the dorsolateral prefrontal cortex (DLPFC) contribute to the synchronization of pyramidal neurons, which is necessary for EF performance. Additionally, given the theory of abnormal synaptic plasticity and excitation/inhibition ratio in ASD, as well as the ability of TMS to modify cortical excitability and plasticity, it leads to exploring the therapeutic potential of rTMS in ASD. This study examines the effectiveness of low-frequency rTMS in improving social, cognitive, and sensory function in individuals with ASD. Further understanding of the effect of low-frequency rTMS in altering the cognitive function in ASD individuals with ASD may help to achieve some answers related to the mechanism behind ASD.

DETAILED DESCRIPTION:
Statement of the Problem:

Autism spectrum disorder (ASD) is a complex neurodevelopmental disorder. Core ASD symptoms include impairments in social communication and restricted and repetitive behaviors, interests, and activities. ASD may also present with secondary signs, including hyperactivity, self-injury, and co-occurrence of some psychiatric conditions, e.g., anxiety and major depression. The symptoms of ASD are persistent and typically appear during the first three years of life. It can be recognized and clinically evident in early childhood.

In most cases, but not all, ASD symptoms might follow a steady course without remission. However, deficits and impairment in social skills and behavioral patterns may not be noticed and diagnosed as symptoms of ASD until the child faces significant life demands such as social, educational, and occupational tasks. Moreover, this functional limitation may vary among persons with ASD and could develop over time.

In the past 50 years, ASD's description has changed from a rare disease of childhood-onset to a well-publicized, advocated, and researched lifelong condition, recognized as relatively common and very heterogeneous. Since the 1970s, several studies have reported increased ASD cases. The report documented that the male/female ratio is approximately 4 per 1. According to the Centers for Disease Control, the prevalence of ASD increased from 1 in 80 (1.25%) in 2011-2013 to 1 in 31 children (3.2%) aged 8 years, and the corresponding figure for the whole of the United States in 2022 was 8 and 9. In the Gulf countries, systematic review studies of the epidemiology of autism revealed a prevalence ranging from 1.4 to 29/10,000 persons. In a study in Taif, Saudi Arabia, the estimated prevalence of autism in primary school children aged 7-12 years was 0.035%. Reviews of the literature have revealed no recent prevalence statistics for children with autism/ASD in Saudi Arabia. The Saudi Ministry of Health has indicated that one in every 160 children has an ASD.

ASDs are a financial, emotional, and social burden. An autistic child's care causes more emotional burden to the parents than that of parents, compared to that of parents taking care of terminally ill children.

Social cognition is a broad term that describes cognitive processes related to perceiving, understanding, and implementing linguistic, auditory, visual, and physical cues that communicate emotional and interpersonal information. It is also defined as the perception of others, the perception of self, and interpersonal knowledge. It's the ability to understand, perceive, and interpret information about others and ourselves in a social context. It includes a wide range of processes that allow people to perceive and interpret rapidly changing social information and respond appropriately to social stimuli quickly, effortlessly, and flexibly. Also, social cognition ability gives meaning to the actions of others.

Assessment of social cognition, primarily focusing on four key domains, such as theory of mind (ToM), emotional empathy, and social perception and behavior, has been increasingly evaluated in clinical settings, given the potential implications of impairments of these skills for therapeutic decision-making. Cognitive impairment is defined as when a person has trouble remembering, learning new things, concentrating, or making decisions that affect their everyday life. The common signs of cognitive impairment may include loss of memory. Asking the same question frequently or repeating the same story over and over, unable to recognize familiar people or places, having trouble exercising judgment, such as knowing what to do in an emergency, changes in mood or behavior, difficulty in vision, difficulty planning or carrying out tasks, such as following a recipe or keeping track of monthly bills.

Studies showed that alterations in social cognition ability were associated with autism, autism severity, and autistic traits. Impairments in social cognition are often highlighted as a potential mechanism underlying social disability in autism spectrum disorder. Different social skills programs have been developed for autistic adults based on the assumption that improving social understanding and ability will improve functional outcomes.

Transcranial magnetic stimulation (TMS) is one method used to deliver electrical stimuli through the scalp in conscious humans. Generally, single-pulse TMS (including paired-pulse TMS) is used to explore brain functioning. In contrast, repetitive TMS (rTMS) is used to induce changes in brain activity that can last beyond the stimulation period. Therefore, TMS and rTMS are indirect and non-invasive methods to induce excitability changes in the motor cortex via a wire coil, generating a magnetic field that passes through the scalp. TMS Non-invasive TMS of the motor cortex leads to a twitch in the target muscle, evoking motor-evoked potential (MEP) on electromyography. As per the literature, TMS might help regulate gamma oscillations, reduce behavioral symptoms, and normalize executive and autonomic dysfunction signs. TMS is a valuable technique for assessing the underlying neurophysiology associated with several neuropathologies. It is a unique tool for establishing potential neural mechanisms responsible for disease progression. Recently, rTMS has been advanced as a potential therapeutic technique to treat selected neurologic disorders. Such neurological disorders include Parkinson's disease, Huntington's disease, amyotrophic lateral sclerosis, and multiple sclerosis.

Moreover, worldwide, multiple studies have repeatedly demonstrated that TMS has antidepressant effects more significantly than sham treatment and that these effects are clinically meaningful. For diagnostic uses, TMS is a potential diagnostic tool in movement disorders. TMS is used worldwide and represents a novel technique with both diagnostic and therapeutic potential. TMS is used to study cortical excitability and intracortical inhibition and investigate cortical and cortico-spinal plasticity mechanisms implicated in ASD pathophysiology. Published studies showing promising results concluded that specific rTMS protocols targeting particular regions of the cortex might lead to improvement in specific behavioral deficits in some individuals with ASD; both the investigative and therapeutic results have been mixed. rTMS and other electrical stimulation devices can modulate the brain's functioning in either a facilitatory or suppressive manner and, when applied over several sessions, can have an additive effect lasting several months. If theories are correct that cortical mechanisms of excitability, connectivity, and plasticity are abnormal in ASD, then rTMS can modulate these mechanisms. Overall, in the hands of trained technicians, rTMS might have great potential as both a diagnostic and therapeutic tool for ASD.

ELIGIBILITY:
Target population:

* Autistic individuals
* previously Diagnosed with ASD using the American Psychiatric Association's DSM-V criteria
* previously Diagnosed using the Autism Diagnostic Observation Schedule (ADOS).

Inclusion Criteria:

* Male and female ASD individuals
* age between 5 and 11 years old
* diagnosed with ASD on prior clinical assessment using the American Psychiatric Association's DSM-V criteria and corroborated by assessment using the Autism Diagnostic Observation Schedule (ADOS).
* Normal hearing ability based on past hearing screens.
* Participation will be limited to higher functioning (intelligence quotient [IQ] >70) to maximize successful completion of tested paradigms, maintain alertness/attention, furthermore, the ability to follow instructions.

Exclusion Criteria:

* Individuals that are known to have epilepsy ( including Hx. of febrile convulsion) or have a family history of epilepsy.
* Any individual with a previous Hx. Of head injuries
* Any individual has been diagnosed with psychiatric illness, including ADHD, depression, psychosis, bipolar disorder, anxiety disorders, or OCD.
* Individuals using a combination of Psychotropic Medications known for their significant seizure threshold lowering potential, for example, and not as a limitation: Bupropion, Citalopram, Duloxetine, Fluoxetine, Fluvoxamine, Mirtazapine, Paroxetine, Sertraline, Venlafaxine, Tricyclics, Olanzapine, Quetiapine, Aripiprazole, Ziprasidone, and Risperidone.
* The presence of metallic objects, e.g., cranium clips or implanted biomedical devices.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Cognitive function | of intervention and 2 week, 3 Months after the last session in intervention for each participant
  Measure the cognitive function by using Cambridge Neuropsychological Test Automated Battery (CANTAB) spatial working memory task, looking of any Statistical significance changes in this score of cognitive testing by using CANTAB battery in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
Severity level of Autism Spectrum disorders (ASD) | pre-intervention and 2 week then 3 Months after the last session in intervention for each participant
  Any Statistical significance change in the severity level of Autism (ASD) , looking for any changes in the score of Childhood Autism Rating Scale,Second Edition (CARS2-ST) in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
  Score will be represented as Total row score and will be interpreted based on the following : for the age between 2-12 years old
  * (15-29.5) Minimal to no symptoms of autism spectrum disorder
  * (30 - 36.5) Mild to moderate symptoms of autism spectrum disorder
  * ( 37 and higher) Severe symptoms of autism spectrum disorder. CARS2-ST Score minimum= 15 and maximum= - , high CARS scores mean a worse outcome.
Autism Spectrum disorder (ASD) Severity level | pre-intervention and 2 week then 3 Months after the last session in intervention for each participant
  Any Statistical significance change in the severity level of Autism (ASD) , looking for any changes in the score of The Social Responsiveness Scale (SRS) teste in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
  Score will be represented as Total T-score and will be interpreted based on the following:
  * T-score of 59T or less ; the result in the normal range.
  * T-score of 60T through 75T; the result in the mild to moderate range.
  * T-score of 76T or higher; The result in the severe range. high SRS T-scores mean a worse outcome.
Blood Biomarker ( Microtubule associated proteins (MAPs) ). | pre-intervention and 2 week then 3 Months after the last session in intervention for each participant
  Any Statistical significance change in the plasma levels of Blood biomarkers in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
  Score will be represented as plasma concentration , Units of Measure: concentration unit pg/ml
Blood Biomarker ( Neuron Specific Enolase (NSE);MYO 16 (myosin XVI); kirre like nephrin family adhesion molecule 3 (KIRREL3) ). | pre-intervention and 2 week then 3 Months after the last session in intervention for each participant
  Any Statistical significance change in the plasma levels of Blood biomarkers in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
  Score will be represented as plasma concentration , Units of Measure: concentration unit ng/ml

SECONDARY OUTCOMES:
Psychology and behaviours | pre-intervention and 2 week then 3 Months after the last session in intervention for each participant
  Any change in Psychology and behaviours in participants , looking for significant statistical analysis in the score of The Child Behavior Checklist (CBCL) in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
  The CBCL uses a normative sample to create standard scores+ Percentile scores. These compare the raw score to what would be typical compared to responses for participants of the same gender and similar age . The standard scores are scaled so that 50 is average for the participants age and gender, with a standard deviation of 10 points. Higher scores indicate greater problems.
Language,Speech and Communication skills | pre-intervention and 2 week then 3 Months after the last session in intervention for each participant
  Any speech and communication skills change in participants , looking for significant statistical analysis in the score of Orion's Pragmatic Language skills in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
  Score will be represented as Total row score for each test Item in scale higher scores mean worse outcome.
Sensory Processing using Sensory Processing Measure (SPM) | Before the beginning of intervention and 2 week, 3 Months after the last session in intervention for each participant
  Any change in participants Sensory Processing , looking for significant statistical analysis in the score of Sensory Processing Measure (SPM)- (Home Form); in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
  Score will be represented as Total row score for scale higher scores mean worse outcome. Scores for each scale fall into one of three interpretive ranges: Typical, Some Problems, or Definite Dysfunction
Sensory Processing | Before the beginning of intervention and 2 week, 3 Months after the last session in intervention for each participant
  Any change in participants Sensory Processing , looking for significant statistical analysis in the score of the Short Sensory Profile in the active rTMS group before and after completion of rTMs sessions and in comparison, with the control group.
  Score will be represented as Total row score for scale higher scores mean a better outcome; Total row score will be interpreted based on the following : (38-141) Define difference (142-154) Probable difference (155-190) typical performance

CONTACTS AND LOCATIONS:
Overall Officials: HAYFA A ALGHABBAN, MD,MSc, Principal Investigator — Department of physiology, collage of Medicine, King Saud University
Locations (1):
- Department of Physiology, Autism Research and Treatment Center (ARTC), King Saud University Medical City (KSUMC)/Collage of Medicine, King Saud University, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis DA, Hashimoto T, Volk DW. Cortical inhibitory neurons and schizophrenia. Nat Rev Neurosci. 2005 Apr;6(4):312-24. doi: 10.1038/nrn1648. PMID 15803162
- [Background] Baruth JM, Casanova MF, El-Baz A, Horrell T, Mathai G, Sears L, Sokhadze E. Low-Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) Modulates Evoked-Gamma Frequency Oscillations in Autism Spectrum Disorder (ASD). J Neurother. 2010 Jul 1;14(3):179-194. doi: 10.1080/10874208.2010.501500. PMID 21116441
- [Background] Oberman LM, Rotenberg A, Pascual-Leone A. Use of transcranial magnetic stimulation in autism spectrum disorders. J Autism Dev Disord. 2015 Feb;45(2):524-36. doi: 10.1007/s10803-013-1960-2. PMID 24127165
- [Background] Regier DA, Kuhl EA, Kupfer DJ. The DSM-5: Classification and criteria changes. World Psychiatry. 2013 Jun;12(2):92-8. doi: 10.1002/wps.20050. PMID 23737408
- [Background] Kaat AJ, Gadow KD, Lecavalier L. Psychiatric symptom impairment in children with autism spectrum disorders. J Abnorm Child Psychol. 2013 Aug;41(6):959-69. doi: 10.1007/s10802-013-9739-7. PMID 23605958
- [Background] Fakhoury M. Autistic spectrum disorders: A review of clinical features, theories and diagnosis. Int J Dev Neurosci. 2015 Jun;43:70-7. doi: 10.1016/j.ijdevneu.2015.04.003. Epub 2015 Apr 8. PMID 25862937
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Blumberg SJ, Bramlett MD, Kogan MD, Schieve LA, Jones JR, Lu MC. Changes in prevalence of parent-reported autism spectrum disorder in school-aged U.S. children: 2007 to 2011-2012. Natl Health Stat Report. 2013 Mar 20;(65):1-11, 1 p following 11. PMID 24988818
- [Background] Charman T, Pickles A, Chandler S, Wing L, Bryson S, Simonoff E, Loucas T, Baird G. Commentary: Effects of diagnostic thresholds and research vs service and administrative diagnosis on autism prevalence. Int J Epidemiol. 2009 Oct;38(5):1234-8; author reply 1243-4. doi: 10.1093/ije/dyp256. Epub 2009 Sep 7. No abstract available. PMID 19737794
- [Background] Samsam M, Ahangari R, Naser SA. Pathophysiology of autism spectrum disorders: revisiting gastrointestinal involvement and immune imbalance. World J Gastroenterol. 2014 Aug 7;20(29):9942-51. doi: 10.3748/wjg.v20.i29.9942. PMID 25110424
- [Background] Amr M, Bu Ali W, Hablas H, Raddad D, El-Mehesh F, El-Gilany AH, Al-Shamy H. Sociodemographic factors in Arab children with Autism Spectrum Disorders. Pan Afr Med J. 2012;13:65. Epub 2012 Nov 26. PMID 23346279
- [Background] Developmental Disabilities Monitoring Network Surveillance Year 2010 Principal Investigators; Centers for Disease Control and Prevention (CDC). Prevalence of autism spectrum disorder among children aged 8 years - autism and developmental disabilities monitoring network, 11 sites, United States, 2010. MMWR Surveill Summ. 2014 Mar 28;63(2):1-21. PMID 24670961
- [Background] Christensen DL, Baio J, Van Naarden Braun K, Bilder D, Charles J, Constantino JN, Daniels J, Durkin MS, Fitzgerald RT, Kurzius-Spencer M, Lee LC, Pettygrove S, Robinson C, Schulz E, Wells C, Wingate MS, Zahorodny W, Yeargin-Allsopp M; Centers for Disease Control and Prevention (CDC). Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years--Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2012. MMWR Surveill Summ. 2016 Apr 1;65(3):1-23. doi: 10.15585/mmwr.ss6503a1. PMID 27031587
- [Background] Salhia HO, Al-Nasser LA, Taher LS, Al-Khathaami AM, El-Metwally AA. Systemic review of the epidemiology of autism in Arab Gulf countries. Neurosciences (Riyadh). 2014 Oct;19(4):291-6. PMID 25274588
- [Background] Inglese MD, Elder JH. Caring for children with autism spectrum disorder. Part I: prevalence, etiology, and core features. J Pediatr Nurs. 2009 Feb;24(1):41-8. doi: 10.1016/j.pedn.2007.12.006. Epub 2008 Jun 13. PMID 19159834
- [Background] Friedman S, Samuelian JC, Lancrenon S, Even C, Chiarelli P. Three-dimensional structure of the Hospital Anxiety and Depression Scale in a large French primary care population suffering from major depression. Psychiatry Res. 2001 Nov 30;104(3):247-57. doi: 10.1016/s0165-1781(01)00309-2. PMID 11728614
- [Background] Beer JS, Ochsner KN. Social cognition: a multi level analysis. Brain Res. 2006 Mar 24;1079(1):98-105. doi: 10.1016/j.brainres.2006.01.002. Epub 2006 Feb 28. PMID 16513097
- [Background] Klomjai W, Katz R, Lackmy-Vallee A. Basic principles of transcranial magnetic stimulation (TMS) and repetitive TMS (rTMS). Ann Phys Rehabil Med. 2015 Sep;58(4):208-213. doi: 10.1016/j.rehab.2015.05.005. Epub 2015 Aug 28. PMID 26319963
- [Background] Casanova MF, Sokhadze EM, Casanova EL, Opris I, Abujadi C, Marcolin MA, Li X. Translational Neuroscience in Autism: From Neuropathology to Transcranial Magnetic Stimulation Therapies. Psychiatr Clin North Am. 2020 Jun;43(2):229-248. doi: 10.1016/j.psc.2020.02.004. Epub 2020 Apr 8. PMID 32439019
- See also: Prevalence and clinical characteristics of autism spectrum disorders in school-age children in Taif- KSA — https://www.bibliomed.org/?mno=32442